CLINICAL TRIAL: NCT00335491
Title: A RENEW Intervention for Elderly Cancer Survivors
Brief Title: Exercise in Improving Mobility and Reducing Fatigue and/or Weakness in Older Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul LaStayo, PT, PhD, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14551; R21CA114523 (NIH); P30CA042014 (NIH); UUMC-R21CA114523; NCT00286715 (obsolete NCT alias)
Record Dates: First submitted 2006-06-08; First posted 2006-06-12 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Bladder Cancer; Breast Cancer; Colorectal Cancer; Esophageal Cancer; Fatigue; Lung Cancer; Lymphoma; Ovarian Cancer; Prostate Cancer
Keywords: small cell lung cancer; non-small cell lung cancer; colon cancer; prostate cancer; breast cancer; male breast cancer; fatigue; lymphoma; ovarian epithelial cancer; bladder cancer; esophageal cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Fatigue; Lung Neoplasms; Lymphoma; Ovarian Neoplasms; Prostatic Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Breast Neoplasms, Male; Carcinoma, Ovarian Epithelial | interventions — Therapeutics; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: exercise intervention — 12 weeks of 3x/week training on a recumbent eccentric stepper
  Other Names: Eccentron
Procedure: complementary or alternative medicine procedure — 12 weeks of 3x/week training on the eccentron
  Other Names: Eccentron
Procedure: fatigue assessment and management — The visual analog scale will be used to assess muscle soreness from the previous exercise session
Procedure: physical therapy — 12 weeks of 3x/week training on the eccentron

SUMMARY:
RATIONALE: Exercise may help improve mobility and relieve fatigue and/or weakness in cancer survivors. It is not yet known whether exercise is more effective than standard therapy in improving mobility and reducing fatigue and/or weakness in older cancer survivors.

PURPOSE: This randomized clinical trial is studying exercise to see how well it works compared to standard therapy in improving mobility and reducing fatigue and/or weakness in older cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the perception of, and the patterns of change in fatigue, weakness, physical activity level, and functional status in elderly cancer survivors who undergo Resistance Exercise via Negative-Eccentric Work (RENEW) vs standard care.
* Compare changes in muscle structure, function (strength + power production and metabolic function) and mobility.
* Evaluate the patient's adherence to and satisfaction with the RENEW intervention.

OUTLINE: This is a prospective, randomized, controlled, longitudinal study. Patients are randomized to 1 of 2 intervention arms.

* Arm I: Patients undergo resistance exercise via negative-eccentric work (RENEW), using a special seated stationary leg exercise machine, 3 times a week for up to 12 weeks. Exercise exertion and duration is gradually increased weekly for the first 4-5 weeks of RENEW.
* Arm II: Patients receive standard care. In both arms, fatigue, weakness, physical activity, functional status, muscle structure and function, and mobility are assessed at baseline and then at 12 weeks after completion of study intervention. Fatigue and weakness are also assessed weekly during study intervention. Patients in arm I also undergo isometric strength assessment weekly during RENEW and assessment of adherence to and satisfaction with RENEW at 12 weeks after completion of RENEW.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Survivor of breast, prostate, colon, lung, lymphoma, ovarian, bladder, or esophageal cancer with no evidence of disease
* At least moderate levels of fatigue and/or weakness
* Impaired mobility but ambulatory and medically able to participate in an exercise regimen

  * No impaired knee flexion, defined as < 90º

PATIENT CHARACTERISTICS:

* Folstein Mini-Mental Status Examination score ≥ 23
* No extreme claustrophobia
* No diagnosed chronic fatigue syndrome/disorder
* No neurological impairments, including the following:

  * Central nervous system disorder (e.g., multiple sclerosis or Parkinson's disease)
  * Neurological insult (cerebrovascular attack) that manifests in a mobility disorder
* No myopathic disease (e.g., focal myopathy) that effects skeletal muscle structure/function
* No rheumatological disease that has an effect on muscle and/or mobility (e.g., polymyalgia rheumatica)

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior regular aerobic or resistance exercise

  * Regular exercise defined as 2-3 times per week
* At least 6 months since prior cancer treatment (surgery, radiation, and/or chemotherapy )
* No concurrent cancer-related treatment other than hormonal therapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Patient perception and pattern of change | 3 months of training followed by 6 and 12 months of no formal training
  To explore the participant's perception and pattern of change in fatigue, weakness, physical activity level and functional status

SECONDARY OUTCOMES:
Structural and function changes | 3 months of training followed by 6 and 12 months of no formal training
  To explore whether changes in muscle structure and function (strength and power production and metabolic function) and mobility occur following twelve weeks of training with RENEW

CONTACTS AND LOCATIONS:
Overall Officials: Paul C. LaStayo, PhD, PT, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] LaStayo PC, Marcus RL, Dibble LE, Smith SB, Beck SL. Eccentric exercise versus usual-care with older cancer survivors: the impact on muscle and mobility--an exploratory pilot study. BMC Geriatr. 2011 Jan 27;11:5. doi: 10.1186/1471-2318-11-5. PMID 21272338